CLINICAL TRIAL: NCT00442845
Title: ACTFAST: Achieve Cholesterol Targets Fast With Atorvastatin Stratified Titration. A Multicenter, Twelve-Week Treatment, Single Step Titration, Open-Label Study Assessing The Percentage Of Dyslipidemic High-Risk Patients Achieving Low Density Lipoprotein Cholesterol (LDL-C) Target With Atorvastatin Starting Doses Of 10 Mg, 20 Mg, 40 Mg, And 80 Mg
Brief Title: Establish The Benefits Of Using Various Starting Doses Of Atorvastatin On Achievement Of Cholesterol Targets (ACTFAST)
Acronym: ACTFAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581087
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronary Arteriosclerosis; Diabetes Mellitus, Type 2; Cerebrovascular Accident; Dyslipidemia; Peripheral Vascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Stroke; Dyslipidemias; Peripheral Vascular Diseases | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin (Lipitor)

SUMMARY:
Physicians tend to always use the lowest dose of statins to initiate therapy even in subjects who require large reductions in cholesterol. The study evaluates if selecting the starting dose based on baseline and target LDL-C cholesterol would provide better results (ie proportion of subjects resching target)

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol blood levels (LDL-cholesterol above 100 mg/dL up to 220 mg/dL.
* Triglycerides up to 600 mg/dL.
* History of coronary artery disease (ex.: heart attack, angina), stroke, diabetes or at high risk of such events

Exclusion Criteria:

* Pregnancy or lactation, use of high statin doses (>40mg) at baseline, liver or renal problems, use of other drugs that would interfere with evaluation of efficacy or cause safety problems, uncontrolled hypertension, diabetes or hypothyroidism, recent cardiac event of procedure, high baseline CPK levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2080
Dates: Start 2003-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a LDL-C target of < 100 mg/dL (2.6 mmol/L) after 12 weeks.

SECONDARY OUTCOMES:
Percentage of subjects achieving:
LDL-C target <100 mg/dL (<2.6 mmol/L) after 6 weeks of treatment.
Total cholesterol (TC)/HDL-C ratio target (<4.0) after 6 and 12 weeks of treatment.
Either the LDL-C <100mg/dL (<2.6 mmol/L) or TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment.
Both the LDL-C <100mg/dL (<2.6 mmol/L) and TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment.
LDL-C <100mg/dL (<2.6 mmol/L) or TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment by LDL-C strata.
LDL-C target (<100 mg/dL) by primary inclusion diagnosis (CHD, CHD-equivalent, diabetes or 10-year CHD risk-equivalent >20%).
The mean percent change in LDL-C, high density lipoprotein cholesterol (HDL-C),TC/HDL-C ratio, non HDL-C (in subjects with triglycerides [TG] ≥200 mg/dL or 2.3 mmol/L), TC and TG from baseline to 6 and 12 weeks of treatment.
Change from baseline in apolipoprotein-B (Apo-B) and change from baseline in glycosylated hemoglobin (HbA1c) was assessed at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (121):
- Pfizer Investigational Site, Mississauga, Ontario, Cameroon
- Canada (55):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Medicine Hat, Alberta
  - Pfizer Investigational Site, Red Deer, Alberta
  - Pfizer Investigational Site, Campbell River, British Columbia
  - Pfizer Investigational Site, Maple Ridge, British Columbia
  - Pfizer Investigational Site, Nanaimo, British Columbia
  - Pfizer Investigational Site, New Westminster, British Columbia
  - Pfizer Investigational Site, Richmond, British Columbia
  - Pfizer Investigational Site, Surrey, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Vernon, British Columbia
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Brandon, Manitoba
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Ajax, Ontario
  - Pfizer Investigational Site, Brampton, Ontario
  - Pfizer Investigational Site, Burlington, Ontario
  - Pfizer Investigational Site, Cambridge, Ontario
  - Pfizer Investigational Site, Cornwall, Ontario
  - Pfizer Investigational Site, Etobicoke, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Niagara Falls, Ontario
  - Pfizer Investigational Site, North YORK, Ontario
  - Pfizer Investigational Site, Orillia, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Rexdale, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Simcoe, Ontario
  - Pfizer Investigational Site, Thunder Bay, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Weston, Ontario
  - Pfizer Investigational Site, Whitby, Ontario
  - Pfizer Investigational Site, Willowdale, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Cowansville, Quebec
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Joliette, Quebec
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Maria, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Newport, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Repentigny, Quebec
  - Pfizer Investigational Site, Saint-Hyacinthe, Quebec
  - Pfizer Investigational Site, Saint-Lambert, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, St-georges (beauce), Quebec
  - Pfizer Investigational Site, Thetford-Mines, Quebec
  - Pfizer Investigational Site, Vaudreuil, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
  - Pfizer Investigational Site, Québec
- Italy (28):
  - Pfizer Investigational Site, Tricase, (LE)
  - Pfizer Investigational Site, Vimercate, (MI)
  - Pfizer Investigational Site, Somma Lombardo, (VA)
  - Pfizer Investigational Site, Asti
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Belluno
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Bolzano
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Chieti
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Foggia
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Novara
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Potenza
  - Pfizer Investigational Site, Prato
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Salerno
  - Pfizer Investigational Site, San Donato Milanese
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Savona
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Venezia
- Spain (13):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Girona, Catalonia
  - Pfizer Investigational Site, Galdakao, Vizcaya
  - Pfizer Investigational Site, Ávila
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Huelva
  - Pfizer Investigational Site, Jerez de la Frontera
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Marbella
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Tarragona
  - Pfizer Investigational Site, Valencia
- United Kingdom (23):
  - Pfizer Investigational Site, Newtonabbey, Belfast
  - Pfizer Investigational Site, Aylesbury, Buckinghamshire
  - Pfizer Investigational Site, Ely, Cambs
  - Pfizer Investigational Site, Peterborough, Cambs
  - Pfizer Investigational Site, Newtonabbey, CO Antrim
  - Pfizer Investigational Site, Hastings, EAST Sussex
  - Pfizer Investigational Site, High Valleyfield, FIFE
  - Pfizer Investigational Site, Rutherglen, Glasgow
  - Pfizer Investigational Site, Leslie, FIFE, Glenrotheshire
  - Pfizer Investigational Site, Sunbury-on-Thames, Middlesex
  - Pfizer Investigational Site, Frome, Somerset
  - Pfizer Investigational Site, Barry, South Glamorgan
  - Pfizer Investigational Site, Doncaster, South Yorkshire
  - Pfizer Investigational Site, Stairfoot, Barnsley, South Yorkshire
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, East Horsley, Surrey
  - Pfizer Investigational Site, Atherstone, Warks
  - Pfizer Investigational Site, Balsall Common, WEST Midlands
  - Pfizer Investigational Site, Pound Hill, Crawley, WEST Sussex
  - Pfizer Investigational Site, Trowbridge, Wiltshire
  - Pfizer Investigational Site, Chippenham, Wilts
  - Pfizer Investigational Site, Sheffield, Yorkshire
  - Pfizer Investigational Site, Bath
- Pfizer Investigational Site

REFERENCES:
- [Derived] Gupta M, Martineau P, Tran T, Despres JP, Gaw A, de Teresa E, Farsang C, Gensini GF, Leiter LA, Blanco-Colio LM, Egido J, Langer A; ACTFAST investigators. Low-density lipoprotein cholesterol and high-sensitivity C-reactive protein lowering with atorvastatin in patients of South Asian compared with European origin: insights from the Achieve Cholesterol Targets Fast with Atorvastatin Stratified Titration (ACTFAST) study. J Clin Pharmacol. 2012 Jun;52(6):850-8. doi: 10.1177/0091270011407196. Epub 2011 May 24. PMID 21610204
- [Derived] Gensini GF, Gori AM, Dilaghi B, Rostagno C, Gaw A, Blanco-Colio LM, de Teresa E, Egido J, Farsang C, Leiter LA, Martineau P, Nozza A, Langer A; Achieve Cholesterol Targets Fast withAtorvastatin Stratified Titration Investigators. Effect of atorvastatin on circulating hsCRP concentrations: a sub-study of the achieve cholesterol targets fast with atorvastatin stratified titration (ACTFAST) study. Int J Cardiol. 2010 Jul 23;142(3):257-64. doi: 10.1016/j.ijcard.2008.12.213. Epub 2009 Feb 12. PMID 19217176
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581087&StudyName=Establish+The+Benefits+Of+Using+Various+Starting+Doses+Of+Atorvastatin+On+Achievement+Of+Cholesterol+Targets+%28ACTFAST%29